CLINICAL TRIAL: NCT05917405
Title: FLUCLORIC: Randomized Multicentric Phase III Study Comparing the Efficacy of 2 Reduced Intensity Conditioning Regimens (Clofarabine/Busulfan vs Fludarabine/Busulfan) in Adults With AML and Eligible to Allogeneic Stem Cell Transplantation
Brief Title: Study Comparing the Efficacy of 2 RIC Regimens (Clofarabine vs Fludarabine) in Adults With AML Eligible to Allo-SCT
Acronym: FLUCLORIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0524
Record Dates: First submitted 2023-05-16; First posted 2023-06-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia in Remission
Keywords: Acute Myeloid Leukemia; Clofarabine; fludarabine; reduced intensity conditioning regimen; allogeneic stem cells transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Busulfan; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: CloB2 arm (Experimental): * 30 mg/m2/day IV clofarabine for 5 days (day-6 to day-2)
  * 3.2mg/kg/day IV busulfan once daily for 2 days (day -5 and -4)
  * ATG (Thymoglobuline®) 2.5 mg/Kg/day IV for 2 consecutive days (day -2 and -1) Corticosteroids may be used in profilaxis
  Interventions: Drug: Busulfan; Drug: ATG; Drug: Clofarabine
- Comparator: FB2A2 arm (Active Comparator): * 30 mg/m2/day IV fludarabine for 5 days (day-6 to day-2)
  * 3.2 mg/kg/day IV busulfan once daily for 2 days (day -5 and -4)
  * ATG (Thymoglobuline®) 2.5 mg/Kg/day IV for 2 consecutive days (day -2 and -1)
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: ATG

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2/day IV fludarabine for 5 days (day-6 to day-2)
  Arms: Comparator: FB2A2 arm
Drug: Busulfan — 130 mg/m2/day IV busulfan once daily for 2 days (day -4 and -3)
Drug: ATG — Thymoglobuline®: 2.5 mg/Kg/day IV for 2 consecutive days (day -2 and -1)
Drug: Clofarabine — 30 mg/m2/day IV clofarabine for 5 days (day-6 to day-2)
  Arms: Experimental: CloB2 arm

SUMMARY:
Relapse remains the main cause of death in patients with myeloid malignancies, especially after an allotransplant. Using drugs with higher anti-leukemic activity as part of the conditioning regimen is one of the strategies to decrease relapse incidence in this population. Retrospective studies have shown that clofarabine can achieve impressive results compared to the use of fludarabine in acute myeloid leukemia (AML) as part of the conditioning regimen. Confirming such results in a prospective manner would definitely establish the CloB2A2 as a superior reduced-intensity conditioning (RIC) regimen compared to the FB2A2 for AML patients.302 AML patients (151 in each arm) in complete remission at transplant will be included with the main objective to demonstrate a significant better 2-year overall survival for CloB2A2 cases (70% vs 55%). A cost-utility analysis and a cost-effectiveness analysis will be also performed as well as an assessment of the quality of life after transplant. Clofarabine will be furnished to all centers. The duration of the study will be 5 years with 3 years of inclusion and 2 years of follow-up for each patient.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years' old

* De novo or secondary AML (according to ELN 2022 classification) in complete cytological remission at time of transplant (bone marrow blast count < 5%) or MDS/LAM with bone marrow blast count ≤ 5%
* Patients in first or second line therapy are allowed
* Patient eligible to a RIC regimen : patients aged ≥ 60 year old or <60 with co-morbidity(ies).
* Patient with a related or an unrelated matched donor
* Graft using only peripheral blood stem cells
* Performance status ECOG 0 - 2
* Who provide their written informed consent
* Previous allograft allowed
* Affiliated with French social security system or beneficiary from such system
* Women must meet one of the following criteria at the time of inclusion:

  * use adequate contraceptive measures as recommended by the CTFG (Recommendations related to contraception and pregnancy testing in clinical trials v1.1; includes injectable implants, dual hormone birth control pills, intrauterine devices, abstinence from sex, or a sterilized partner), and have a negative pregnancy test (urine or serum pregnancy test) prior to receiving the first dose of study drug;
  * or be post-menopausal (over 50 years of age with amenorrhea for at least 12 months after discontinuation of all exogenous hormonal therapy)
  * or (if under 50 years of age) have been amenorrheic for at least 12 months after discontinuation of exogenous hormonal therapy and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels corresponding to post-menopausal levels
  * or have undergone irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (this operation must be documented).
  * Contraception methods must be prescribed using effective contraceptive methods during treatment and within 6 months for women of childbearing age (WOCB) and 6 months for men in case they have sexual relations with WOCB after the last dose of Fludarabine/Clofarabine.

Exclusion Criteria:

* Pro-myelocytic leukemia
* Patient eligible to a myeloablative conditioning regimen
* Patient with haploidentical, mismatched unrelated donor or umbilical cord blood
* Pregnant or breastfeeding woman or patient refusing contraceptive mesures
* HIV positive
* Active Hepatitis B or C
* Left ventricular ejection fraction < 50%.
* DLCOc <40%
* Uncontrolled infection
* Uncontrolled haemolytic anaemia
* Creatinine clearance < 50 ml/min (evaluated by MDRD or CKDEPI).
* Serum bilirubine > 30 mmol/l, Cytolysis > 5 the upper limit range
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 2 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation to another interventional study during the last month or expected participation to another interventional study during participation to the FLUCLORIC study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2028-09-14 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
To compare 2-year OS between patients with AML in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT. | 2 years
  OS is defined as the time from day 1 of conditioning to death or last follow-up for survivors.

SECONDARY OUTCOMES:
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT: Engraftment, primary and secondary graft failure | day +30/42 and 2 years
  * Engraftment: PNN >500/mm3 + donor chimerism >=5% (day +30/42)
  * Primary and secondary graft failure: donor chimerism <5% at day +30/42 post-transplant (primary) or at distance of transplant after achieving engraftment (secondary)
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT: Neutrophils and platelet recoveries | 2 years
  * Neutrophils recovery: the first of three consecutive days with neutrophils ≥500/mm3 after aplasia from day 0 of the graft
  * Platelets recovery: the first of three consecutive days with platelets ≥20000/mm3 without transfusion after aplasia from day 0 of the graft
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT: 2-year DFS | 2 years
  DFS: time from day1 of the conditioning to time without death or evidence of relapse or disease progression censored at the date of last follow-up.
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT:-2-year relapse incidence | 2 years
  Relapse: any event related to progression or re-occurrence of the disease from day 1 of the conditioning.
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT:2-year NRM | 2 years
  NRM: death from any cause without previous relapse or progression from day 1 of the conditioning
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT:Incidence of acute and chronic graft versus host disease (GVHD) | Day 90 and 2 years
  * Acute GVHD: NIH criteria
  * Chronic GVHD: NIH criteria
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo-SCT:Incidence of GVHD free relapse free survival (GRFS) | 2 years
  GRFS: alive with no previous grade III-IV acute GvHD, no moderate or severe chronic GvHD and no relapse from day 1 of the conditioning
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo SCT:Chimerism | days +30, +60, +90
  Chimerism: peripheral blood and CD3 T cells by molecular markers at days +30, +60, +90/100
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo- SCT:Immune reconstitution | 3, 6 and 12 months
  Immune reconstitution: Immunophenotype of PB lymphocytes and EPP: CD4, CD8, B, NK, EPP at 3, 6 and 12 months
To compare between AML patients in complete remission receiving either a CloB2A2 or a FB2A2 RIC regimen for allo- SCT: Minimal residual disease (MRD) | days +30 and +90
  Minimal residual disease (MRD): before transplant, at day +30 and day +90/100 by flow cytometry, molecular biology and NGS (if available) (ELN 2022 recommendation, Dohner et al Blood 2022)
Comparison of infections after FB2A2 vs CloB2A2: bacterial, viral, parasitic and fungal | day+90
  Comparison of infections after FB2A2 vs CloB2A2: bacterial, viral, parasitic and fungal between day 0 and day+90/100
Quality of life using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) | Days -7, +30, +90, +180, +360 and +720
  Score of the QLQ-C30 questionnaire, including 30 questions assessing some aspects of the quality of life of cancer patients. The total score ranges from 0 to 100.
Quality of life using the and FACT-BMT (Functional Assessment of Cancer Therapy - Bone Marrow Transplant)) | Days -7, +30, +90, +180 and +360
  Score of the FACT-BMT questionnaire, including 50 questions assessing some aspects of the quality of life of cancer patients. The total score ranges from 0 to 200.
comparison of the cost of graft hospitalization between the 2 arms | 2 years
  Graft hospitalization cost: Comparison between both groups in terms of length of stay (in days), use of antibiotics (type and length in days)
comparison of the cost of graft hospitalization between the 2 arms | 2 years
  Graft hospitalization cost: Comparison between both groups in terms of blood products administered (numbers)
health benefit measurement in both treatment arms | Days -7, +30, +90, +180, +360 and +720.
  General Health State with Euroqol EQ-5D-5L questionnaire at Days -7, 30, 90, 180, 360 and 720; 5 answers are possible.
Evaluation of economic efficiency of a CloB2A2 compared to a FB2A2 RIC regimen for allo-SCT, from a collective perspective (considering costs to the National Health Insurance system, hospital and patients)with a 24-month time horizon. | 2 years
  Health Economic study: Incremental cost-utility ratio (ICUR, cost per quality-adjusted life year [QALY] gained) and incremental cost-effectiveness ratio (ICER, cost per life year gained), from a collective perspective and with a 24-month time horizon
Comparison of Overall survival (OS) between patients in first vs second line therapy and impact of clofarabine vs fludarabine in each sub-group. | 2 years
  Comparison of time from D1 of conditioning to death or last follow-up for survivors
Comparison of DFS between patients in first vs second line therapy and impact of clofarabine vs fludarabine in each sub-group. | 2 years
  Comparison of time from day1 of the conditioning to time without death or evidence of relapse or disease progression censored at the date of last follow-up.
Comparison of Overall survival (OS) between patients receiving a first vs a second allograft and impact of clofarabine vs fludarabine in each sub-group. | 2 years
  Comparison of time from D1 of conditioning to death or last follow-up for survivors
Comparison of DFS between patients receiving a first vs a second allograft and impact of clofarabine vs fludarabine in each sub-group. | 2 years
  Comparison of time from day1 of the conditioning to time without death or evidence of relapse or disease progression censored at the date of last follow-up.
Comparison of occurence of Veno-occlusive disease between patients receiving clofarabine vs fludarabine.n day 0 and day+90/100 | day+90
  Comparison of occurrence of veno-occlusive disease : (Mohty et al, BMT 2016) betwee
Safety assessment | 2 years
  Safety assessment: the safety assessment shall be done by collecting all adverse events that occur during the research. All adverse event (except GvHD) shall be graded according to CTC-AE Toxicity Grading Scale (version 5).

CONTACTS AND LOCATIONS:
Overall Officials: patrice CHEVALLIER, Pr, Principal Investigator — Nantes University Hospital
Locations (23):
- France (23):
  - CHU de Nantes, Nantes, Loire Atlantique
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CRLC Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - APHP Créteil, Créteil
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Paris St-Louis, Paris
  - Pitie-Salpetriere, APHP, Paris
  - St-Antoine, APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU St-Etienne, Saint-Etienne
  - CRLC Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No